CLINICAL TRIAL: NCT07241312
Title: Investigation of the Relationship Between Muscle Oxygenation and Upper Extremity Exercise Capacity, Respiratory and Peripheral Muscle Strength, and Activities of Daily Living in Patients With Chronic Neck Pain
Brief Title: Relationship Between Muscle Oxygenation and Upper Extremity Exercise Capacity in Patients With Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Ph.D, Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU530
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Neck Pain
Keywords: chronic neck pain; upper extremity; muscle oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Neck Pain Group: Individuals between the ages of 18-65 who have had neck pain for at least 12 weeks, who were followed up in the Physical Therapy Outpatient Clinic of the Department of Physical Medicine and Rehabilitation will be included in the study.

SUMMARY:
The aim of the study was to investigate the relationship between upper extremity exercise capacity and muscle oxygenation, muscle strength, and activities of daily living in patients with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is an important public health problem that causes disability worldwide Chronic neck pain is defined as the presence of pain in an individual's neck area for more than twelve weeks. Chronic neck pain negatively affects the daily living activities of the individual; functional limitation causes job loss.

Neck pain has been observed to be associated with the trapezius muscle and impaired microcirculation in the trapezius muscle and inadequate muscle blood flow and oxygenation.

In addition, neck pain has been stated to reduce upper extremity performance. However, most of the results regarding the relationship between muscle activity and pain are not consistent. In addition, there are studies showing that respiratory muscles as well as peripheral muscles are affected in these patients. In the light of all this information, it was concluded that there may be a relationship between upper extremity exercise capacity and the oxygen level of the trapezius muscle and activities of daily living in patients with chronic neck pain. In this context, the aim of the study was to investigate the relationship between upper extremity exercise capacity and muscle oxygenation, muscle strength and activities of daily living in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neck pain lasting at least 3 months due to one of the following problems: cervical strain or sprain, cervical disc lesions, cervical spondylosis, facet joint dysfunction, and myofascial pain syndrome.

Exclusion Criteria:

* Neck pain intensity during activity is below 3 points according to the Visual Analog Scale
* Upper extremity motor deficit on neurological examination
* Any surgery related to neck problems
* Cervical radiculopathy
* Any upper extremity surgery
* Any rheumatic and/or neurological disease or any disease affecting the vestibular system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 who have had neck pain for at least 12 weeks, who were followed up in the Physical Therapy Outpatient Clinic of the Department of Physical Medicine and Rehabilitation will be included in the study.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-11-24 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Trapezius Muscle Oxygen Saturation | Day 1
  Patients' trapezius muscle oxygen saturation will be measured using a near infrared spectroscopy (Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA)).
Evaluation of upper extremity capacity | Day 1
  Patients' upper extremity functional exercise capacity will be evaluated with six-minute pegboard and ring test.

SECONDARY OUTCOMES:
Evaluation of peripheral muscle strength | Day 2
  Patients' shoulder abductor and shoulder flexor, elbow flexor and upper trapezius muscle strength will be evaluated with a portable hand dynamometer (KFORCE Muscle Controller®, KinventTM, France).
Evaluation of respiratory muscle strength | Day 2
  An electronic mouth pressure device in accordance with American Thoracic Society and European Respiratory Society criteria will be used to evaluate respiratory muscle strength (Micro Medical MicroRM, UK).
Evaluation of activity of daily living | Day 2
  The Glittre activity of daily living test will be used to evaluate patients' activities of daily living.
Evaluation of upper extremity functional status | Day 1
  Upper Extremity Functional Index will be used to evaluate the upper extremity functional status of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No